CLINICAL TRIAL: NCT01904058
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate LUM001, an Apical Sodium-dependent Bile Acid Transporter Inhibitor (ASBTi) in Combination With Ursodeoxycholic Acid (UDCA) in Patients With Primary Biliary Cirrhosis
Brief Title: Phase 2 Study to Evaluate LUM001 in Combination With Ursodeoxycholic Acid in Patients With Primary Biliary Cirrhosis
Acronym: CLARITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUM001-201; 2013-000482-36 (EudraCT Number)
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: PBC; Primary Biliary Cirrhosis
Keywords: PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LUM001 and Ursodeoxycholic Acid (UDCA) (Experimental): Administered orally once daily
  Interventions: Drug: LUM001; Drug: Ursodeoxycholic Acid
- Placebo and Ursodeoxycholic Acid (UDCA) (Placebo Comparator): Administered orally once daily
  Interventions: Drug: Placebo; Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: LUM001
  Arms: LUM001 and Ursodeoxycholic Acid (UDCA)
Drug: Placebo
  Arms: Placebo and Ursodeoxycholic Acid (UDCA)
Drug: Ursodeoxycholic Acid
  Other Names: UDCA

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, multicenter study. It is a 13-week Phase 2 study in adults with primary biliary cirrhosis designed to compare the effect of daily dosing with UDCA in combination with LUM001 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Primary Biliary Cirrhosis
2. Moderate to severe pruritus
3. Taking ursodeoxycholic acid (UDCA) for at least 6 months, or unable to tolerate UDCA
4. Ability to understand and willingness to sign informed consent prior to initiation of any study procedures

Exclusion Criteria:

1. History or presence of other concomitant significant liver disease
2. Liver transplant
3. Known HIV infection
4. Women who are pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (24):
- United States (17):
  - Scripps Clinic, La Jolla, California
  - University of California at Davis, Sacramento, California
  - University of Miami, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Gastroenterology, Saint Paul, Minnesota
  - St. Louis University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Advanced Liver Therapies at St. Lukes Episcopal Hospital, Houston, Texas
  - University of Utah Health Science Center, Salt Lake City, Utah
  - Liver Institute of Virginia, Newport News, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - University of Washington Harborview Medical Center, Seattle, Washington
- University Health Network, Toronto Western Hospital, Toronto, Ontario, Canada
- United Kingdom (6):
  - University of Birmingham, Birmingham, England
  - Royal Liverpool & Broadgreen University Hospital, Liverpool, England
  - Newcastle University, Newcastle upon Tyne, England
  - Oxford University Hospitals (John Radcliffe), Oxford, England
  - Royal Free Hospital, London
  - Imperial College London St Mary's Hospital, London

REFERENCES:
- See also: Related Info — http://www.lumenapharma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 24 centers in the United Kingdom, Canada, and the United States between 19 August 2013 and 09 April 2015.
Pre-assignment Details: A total of 87 participants were screened out of which 66 participants were randomized into the study and the remaining 21 were screen failures.
Groups:
- LUM001 10 mg + UDCA (Cohort A): In Cohort A, participants received LUM001 tablet in combination with ursodeoxycholic acid (UDCA) orally once daily at a dosage of 2.5 up to a maximum of 10 milligram (mg) during the dose-escalation period over a 3 week period. Thereafter, participants received LUM001 10 mg tablet along with one placebo matched to LUM001 orally once daily for another 10 weeks, in combination with UDCA. Participants continued UDCA alone for an additional period of 4 weeks.
- LUM001 20 mg + UDCA (Cohort B): In Cohort B, participants received LUM001 tablets in combination with UDCA orally once daily at a dosage of 2.5 mg up to a maximum of 20 mg during the dose-escalation period over a 4 week period. Thereafter, participants received LUM001 20 mg (2x10 mg) tablet orally once daily for another 9 weeks, in combination with UDCA. Participants continued UDCA alone for an additional period of 4 weeks.
- Placebo + UDCA (Cohort A): In Cohort A, participants received placebo (matched to LUM001) once daily for a period of 13 weeks, in combination with UDCA. Participants continued UDCA alone for an additional period of 4 weeks.
- Placebo + UDCA (Cohort B): In Cohort B, participants received placebo (matched to LUM001) for a period of 13 weeks, in combination with UDCA. Participants continued UDCA alone for an additional period of 4 weeks.
Period: Overall Study
Arm/Group | LUM001 10 mg + UDCA (Cohort A) | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B)
Started | 21 | 21 | 11 | 13
Completed | 18 | 21 | 10 | 12
Not Completed | 3 | 0 | 1 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LUM001 10 mg + UDCA (Cohort A) | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B) | Total
Number analyzed (Participants) | 21 | 21 | 11 | 13 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.74) | 53.5 (10.53) | 47.5 (8.14) | 55.8 (8.73) | 53.3 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 11 | 12 | 60
  Male | 1 | 4 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pruritus Using Adult Itch Reported Outcome (ItchRO) Weekly Sum Score at Week 13/ Early Termination (ET)
Description: Pruritus was assessed using ItchRO measure, administered as an electronic diary (eDiary) which was completed by the participants twice daily (morning and evening). (ItchRO) scores ranged from 0 to 10, with 0 representing no itch and 10 representing very severe itching. The highest score between the morning and evening ItchRO reports represented the daily score: a measure of the worst itching over the previous 24-hour period. The weekly sum score was calculated as the sum of the daily scores for the 7 days prior to the time point being reported: 7 days prior to randomization or 7 days prior to Week 13/ET visit.
Time Frame: Baseline and Week 13/ET
Population: The mITT population included all participants who were randomized, received at least 1 dose of treatment, and had at least 1 post-baseline ItchRO assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LUM001 10 mg + UDCA (Cohort A: In Cohort A, participants received LUM001 tablet in combination with ursodeoxycholic acid (UDCA) orally once daily at a dosage of 2.5 up to a maximum of 10 milligram (mg) during the dose-escalation period over a 3 week period. Thereafter, participants received LUM001 10 mg tablet along with one placebo matched to LUM001 orally once daily for another 10 weeks, in combination with UDCA. Participants continued UDCA alone for an additional period of 4 weeks.
Arm/Group | LUM001 10 mg + UDCA (Cohort A | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B)
Number analyzed (Participants) | 21 | 21 | 11 | 13
units on a scale
  Baseline | 48.11 (13.363) | 52.10 (13.780) | 54.64 (9.157) | 49.46 (14.110)
  Change at Week 13/ET | -24.59 (15.240) | -27.67 (19.888) | -26.18 (18.313) | -22.77 (17.123)
Statistical Analysis 1: Comparison: LUM001 10 mg + UDCA (Cohort A vs Placebo + UDCA (Cohort A) vs Placebo + UDCA (Cohort B); The difference between treatment groups in change from Baseline to Week 13/ET in ItchRO weekly sum score evaluated by analysis of covariance (ANCOVA) using generalized linear model (GLM). The model included terms for treatment group, alkaline phosphatase (ALP) level (strata), treatment group by ALP level interaction and Baseline ItchRO weekly sum score as a covariate. Least squares mean change from Baseline to Week 13/ET, along with 95 percentage (%) confidence interval for mean were presented; Test type: Superiority or Other; p = 0.6603, ANCOVA — p-value (LUM001 LS Mean = Placebo LS Mean); Least squares mean difference = -2.28, 95% CI 2-sided [-12.59 to 8.03]
Statistical Analysis 2: Comparison: LUM001 20 mg + UDCA (Cohort B) vs Placebo + UDCA (Cohort A) vs Placebo + UDCA (Cohort B); The difference between treatment groups in change from Baseline to Week 13/ET in ItchRO weekly sum score was evaluated by ANCOVA using a GLM. The model included terms for treatment group, ALP level (strata), treatment group by ALP level interaction, and Baseline ItchRO weekly sum score as a covariate. Least squares mean change from Baseline to Week 13/ET, along with 95% confidence interval for the mean, were presented; Test type: Superiority or Other; p = 0.4380, ANCOVA — p-value (LUM001 LS Mean = Placebo LS Mean); Least squares mean difference = -3.99, 95% CI 2-sided [-14.20 to 6.23]

2. Secondary Outcome: Change From Baseline in Pruritus Using Adult ItchRO Weekly Sum Scores at Weeks 4, 8 and 13
Description: ItchRO scores had a range from 0 to 10, with 0 representing no itch and 10 representing very severe itching. The highest score between the morning and evening ItchRO reports represented the daily score: a measure of the worst itching over the previous 24-hour period. The weekly sum score was calculated as the sum of the daily scores for the 7 days prior to the time point being reported: 7 days prior to randomization or 7 days prior to Week 13/ET visit.
Time Frame: Baseline, Weeks 4, 8 and 13
Population: mITT Population. Here, "n" signifies the number of participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LUM001 10 mg + UDCA (Cohort A) | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B)
Number analyzed (Participants) | 21 | 21 | 11 | 13
units on a scale
  Baseline (n=21, 21, 11, 13) | 48.11 (13.363) | 52.10 (13.780) | 54.64 (9.157) | 49.46 (14.110)
  Change at Week 4 (n=20, 21, 11, 13) | -15.62 (13.708) | -22.19 (18.101) | -10.55 (11.103) | -16.23 (12.749)
  Change at Week 8 (n=20, 21, 10, 13) | -21.92 (13.089) | -23.97 (20.398) | -23.50 (18.585) | -19.15 (15.302)
  Change at Week 13 (n=18, 21, 10, 12) | -27.41 (14.346) | -27.67 (19.888) | -28.50 (17.520) | -22.92 (17.876)

3. Secondary Outcome: Change From Baseline in Pruritus Using Adult ItchRO Average Daily Scores at Weeks 4, 8, 13, and Last Post-baseline Visit (Week 13/ET)
Description: ItchRO scores had a range from 0 to 10, with 0 representing no itch and 10 representing very severe itching. The highest score between the morning and evening ItchRO reports represented the daily score: a measure of the worst itching over the previous 24-hour period. Adult ItchRO average daily score was the sum of daily scores divided by the number of days adult ItchRO was completed, using the 7 days prior to the reported visit date.
Time Frame: Baseline, Weeks 4, 8, 13 and Last Post-baseline visit (Week 13/ET)
Population: mITT Population. Here, "n" signifies the number of participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LUM001 10 mg + UDCA (Cohort A) | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B)
Number analyzed (Participants) | 21 | 21 | 11 | 13
units on a scale
  Baseline (n=21, 21, 11, 13) | 6.873 (1.9091) | 7.442 (1.9686) | 7.805 (1.3082) | 7.066 (2.0158)
  Change at Week 4 (n=20, 21, 11, 13 | -2.231 (1.9587) | -3.170 (2.5859) | -1.506 (1.5861) | -2.319 (1.8212)
  Change at Week 8 (n=20, 21, 10, 13) | -3.131 (1.8703) | -3.424 (2.9139) | -3.357 (2.6549) | -2.736 (2.1860)
  Change at Week 13 (n=18, 21, 10, 12) | -3.915 (2.0496) | -3.952 (2.8411) | -4.071 (2.5028) | -3.274 (2.5537)
  Change at Week 13/ET (n=21, 21, 11, 13) | -3.512 (2.1774) | -3.952 (2.8411) | -3.740 (2.6161) | -3.253 (2.4461)

4. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP) at Weeks 4, 8, 13, and Last Post-baseline Visit (Week 13/ET)
Description: Laboratory serum ALP enzyme levels were evaluated using blood samples collected.
Time Frame: Baseline, Weeks 4, 8, 13 and Last Post-baseline (Week 13/ET)
Population: mITT Population. Here, "n" signifies the number of participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | LUM001 10 mg + UDCA (Cohort A) | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B)
Number analyzed (Participants) | 21 | 21 | 11 | 13
units per liter (U/L)
  Baseline (n=21, 21, 11, 13) | 288.2 (193.91) | 257.6 (190.38) | 253.9 (96.83) | 274.2 (190.85)
  Change at Week 4 (n=20, 21, 10, 13) | -22.1 (54.94) | 13.2 (47.76) | 20.3 (49.68) | -0.7 (39.69)
  Change at Week 8 (n=20, 21, 10, 12 | 2.6 (53.95) | 1.1 (41.98) | 8.8 (38.72) | -4.8 (55.70)
  Change at Week 13 (n=17, 20, 10, 12) | -15.2 (97.19) | 18.5 (56.21) | 24.3 (76.48) | -7.2 (83.70)
  Change at Week 13/ET (n=21, 21, 11, 13) | -8.0 (93.02) | 16.4 (55.60) | 22.9 (72.70) | -7.9 (80.19)

5. Secondary Outcome: Change From Baseline in 5-D Itch Score at Weeks 4, 8, 13, and Last Post -Baseline Visit (Week 13/ET)
Description: The 5-D itch (validated instrument to measure pruritus) scale was developed for the multidimensional quantification of pruritus that is sensitive to change over time. The 5-D itch scale included 5 domains (duration, degree, direction, disability, and distribution of pruritus). The total 5-D score was obtained by scoring each of the domains separately and then summing them together. 5-D total scores ranged between 5 (no pruritus) and 25 (most severe pruritus).
Time Frame: Baseline, Weeks 4, 8, 13 and Last Post-baseline visit (Week 13/ET)
Population: mITT Population. Here, "n" signifies the number of participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo + UDCA (Cohort B: In Cohort B, participants received placebo (matched to LUM001) for a period of 13 weeks, in combination with UDCA. Participants continued UDCA alone for an additional period of 4 weeks.
Arm/Group | LUM001 10 mg + UDCA (Cohort A) | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B
Number analyzed (Participants) | 21 | 21 | 11 | 13
units on a scale
  Baseline (n=21, 21, 11, 13) | 18.7 (3.47) | 19.4 (3.49) | 19.6 (2.94) | 19.2 (3.32)
  Change at Week 4 (n=20, 21, 10, 13) | -4.8 (3.91) | -6.3 (4.96) | -3.4 (3.89) | -4.2 (3.81)
  Change at Week 8 (n=20, 21, 10, 12) | -6.8 (3.16) | -5.9 (5.62) | -6.4 (6.20) | -4.4 (4.27)
  Change at Week 13 (n=18, 21, 10, 12) | -7.4 (3.68) | -7.0 (5.89) | -7.8 (5.94) | -6.1 (4.68)
  Change at Week 13/ET (n=21, 21, 10, 13) | -6.5 (4.11) | -7.0 (5.89) | -7.8 (5.94) | -5.6 (4.79)

6. Secondary Outcome: Change From Baseline in Fasting Serum Bile Acid Level at Weeks 4, 8, 13, and Last Post -Baseline Visit (Week 13/ET)
Description: Laboratory serum bile acid level levels were evaluated using blood samples collected.
Time Frame: Baseline, Weeks 4, 8, 13 and Last Post-baseline visit (Week 13/ET)
Population: mITT Population. Here, "n" signifies the number of participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | LUM001 10 mg + UDCA (Cohort A) | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B)
Number analyzed (Participants) | 21 | 21 | 11 | 13
micromoles per liter
  Baseline (n=21, 21, 11, 13) | 33.110 (30.5943) | 52.460 (94.3892) | 52.615 (64.6162) | 58.434 (73.9895)
  Change at Week 4 (n=20, 21, 10, 13) | -11.204 (31.6132) | -14.465 (58.5891) | -10.221 (50.0398) | 14.317 (75.1092)
  Change at Week 8 (n=20, 21, 10, 12) | -3.968 (45.7388) | -21.983 (78.6134) | -3.585 (52.4398) | 34.893 (67.7189)
  Change at Week 13 (n=18, 21, 10, 12) | -8.122 (48.1290) | -19.098 (81.8452) | 11.481 (44.0465) | 4.123 (46.2170)
  Change at Week 13/ET (n=21, 21, 10, 13) | -4.504 (45.7595) | -19.098 (81.8452) | 11.481 (44.0465) | 3.690 (44.2770)

7. Secondary Outcome: Change From Baseline in Bile Acid Synthesis as Measured by Serum 7 Alpha-Hydroxy-4-Cholesten-3-One C4 Level [7 Alpha C4]) at Weeks 4, 8, 13, and Last Post -Baseline Visit (Week 13/ET)
Description: C4 7 alpha-hydroxy-4-cholesten-3-one is an intermediate in the biochemical synthesis of bile acids from cholesterol and its concentrations reflect the activity of the bile acid synthetic pathway. Elevated levels of C4 indicate bile acid malabsorption. Laboratory C4 levels were evaluated using blood samples collected.
Time Frame: Baseline, Weeks 4, 8, 13 and Last Post-baseline Visit (Week 13/ET)
Population: mITT Population. Here, "n" signifies the number of participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | LUM001 10 mg + UDCA (Cohort A) | LUM001 20 mg + UDCA (Cohort B) | Placebo + UDCA (Cohort A) | Placebo + UDCA (Cohort B)
Number analyzed (Participants) | 21 | 21 | 11 | 13
nanogram per milliliter (ng/mL)
  Baseline (n=21, 21, 10, 13) | 18.74 (16.180) | 13.17 (11.851) | 22.31 (20.769) | 16.98 (33.093)
  Change at Week 4 (n=20, 21, 9, 13) | 8.66 (23.422) | 17.03 (18.380) | -6.80 (6.783) | -0.19 (8.856)
  Change at Week 8 (n=20, 21, 9, 12) | 13.04 (17.895) | 15.03 (31.120) | -12.57 (14.630) | 3.43 (16.666)
  Change at Week 13 (n=18, 21, 9, 12) | 24.38 (38.105) | 6.62 (10.116) | -12.72 (10.374) | 4.56 (13.610)
  Change at Week 13/ET (n=21, 21, 9, 13) | 20.56 (37.312) | 6.62 (10.116) | -12.72 (10.374) | 4.74 (13.047)

8. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the product. A serious adverse event (SAE) was defined as an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly or birth defect; an important medical event that did not meet any of the above criteria but jeopardized the participant or required medical or surgical intervention to prevent one of the outcomes listed above. A TEAE was defined as any AE that occurred during the study, from the start of investigational product dosing through the end of the study (13 weeks of treatment period (or ET) + 14 days ]), or that worsened since the start of dosing.
Time Frame: From the first dose of study drug until the 13 weeks of treatment period (or ET) + 14 days (approximately 15 weeks)
Population: The Safety Population included all participants who were randomized and received at least 1 dose of the study drug. One participant was randomized to LUM001 10 mg, but was down-titrated to 5 mg dose due to tolerability issues. The safety data has been summarized based on the study dose actually received by the participant.
Measure: Number; unit: participants
Groups:
- LUM001 5 mg + UDCA: Participants received LUM001 5 milligram (mg) tablet orally once daily for a period of 13 weeks in combination with UDCA.
- LUM001 10 mg + UDCA: Participants received LUM001 10 mg tablet orally once daily for a period of 13 weeks in combination with UDCA.
- LUM001 20 mg + UDCA: Participants received LUM001 20 mg (2x 10 mg) tablet for 20 mg daily dose in combination with UDCA orally once daily for a period of 13 weeks.
- Placebo + UDCA: Participants received placebo matched to LUM001 tablet orally once daily for a period of 13 weeks in combination with UDCA.
Arm/Group | LUM001 5 mg + UDCA | LUM001 10 mg + UDCA | LUM001 20 mg + UDCA | Placebo + UDCA
Number analyzed (Participants) | 1 | 20 | 21 | 24
participants
  TEAEs | 1 | 19 | 21 | 17
  TESAEs | 0 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until the 13 weeks of treatment period (or ET) + 14 days (approximately 15 weeks)
Description: One subject was randomized to LUM001 10 mg, but was down-titrated to 5mg dose due to tolerability issues. One participant was randomized to LUM001 10 mg, but was down-titrated to 5 mg dose due to tolerability issues. The safety data has been summarized based on the study dose actually received by the participant.
Groups:
- LUM001 5 mg + UDCA: Participants received LUM001 5 mg tablet orally once daily for a period of 13 weeks in combination with UDCA.
Arm/Group | LUM001 5 mg + UDCA | LUM001 10 mg + UDCA | LUM001 20 mg + UDCA | Placebo + UDCA
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/20 | 1/21 | 0/24
Other Adverse Events (participants affected / at risk) | 1/1 | 18/20 | 20/21 | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUM001 5 mg + UDCA (N=1) | LUM001 10 mg + UDCA (N=20) | LUM001 20 mg + UDCA (N=21) | Placebo + UDCA (N=24)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUM001 5 mg + UDCA (N=1) | LUM001 10 mg + UDCA (N=20) | LUM001 20 mg + UDCA (N=21) | Placebo + UDCA (N=24)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (4)
Abdominal Pain (Gastrointestinal disorders) | 1 (3) | 4 (4) | 5 (6) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 4 (6) | 6 (9) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 14 (16) | 11 (19) | 6 (7)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Faeces Discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 5 (6) | 4 (5) | 4 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anal Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 8 (10)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Sinus Operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.